CLINICAL TRIAL: NCT00215592
Title: An Open Label Study Of Zonegran (Zonisamide) In Patients With Partial Onset Seizures
Brief Title: Open Label, Zonegran (Zonisamide) In Partial Onset Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2090-E044-401; 2005-001982-33 (EudraCT Number)
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide

INTERVENTIONS:
Drug: Zonegran

SUMMARY:
To determine the efficacy and safety of adjunctive open label Zonegran treatment in patients with refractory partial seizures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-75.
2. Able and willing to give written informed consent in accordance with the ICH GCP Guidelines.
3. Female subjects of childbearing potential must not be pregnant (as confirmed by negative serum βHCG at screening and negative urine pregnancy test at baseline/during the study), must not be lactating and must use a medically acceptable form of contraception during the study and for at least 1 month after discontinuation of study drug. Medically acceptable contraception as defined here is the oral contraceptive pill, surgical sterilization or hormonal intrauterine device in place for at least 3 months. Women who are less than 2 years post-menopausal are considered to be of childbearing potential.
4. Focal epilepsy, with simple and/or complex partial seizures with or without secondary generalized seizures as defined by the ILAE criteria.
5. Patients with a minimum of 4 partial seizures in the 8 weeks preceding the baseline visit as adequately recorded using a seizure diary card.
6. Patients should be receiving at least 1 but no more than 2 other AEDs as concomitant medication, and the dosage should be stable for at least 8 weeks before the baseline visit.

Exclusion Criteria:

1. History of status epilepticus within the last 5 years.
2. Patients with known significantly impaired renal function and/or severe hepatic impairment to the extent that the protocol dose titration schedule cannot be followed. Note Investigators should consult included SmPC as a guide.
3. Patients suffering from clinically significant psychiatric illness, psychological or behavioral problems which could interfere with study participation.
4. Patients with a history (within the last 12 months) of alcohol or drug abuse or dependency.
5. Patient suffering from any CNS progressive disease that may confound study interpretation, any active CNS infection, demyelinating disease or degenerative neurological disease.
6. Patients with a significant drug sensitivity or significant allergic reaction to any drug including sulfonamides.
7. Subjects considered by the Investigator to be an unsuitable candidate for receiving Zonegran or considered unlikely to comply with the protocol.
8. Any patient contraindicated for Zonegran treatment as per attached SmPC.
9. Any patient who is pregnant and/or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2005-10; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Seizure frequency, compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tone Bjaaland, Study Director — Eisai Limited
Locations (33):
- Universitatsklinikum fur Neurologie, Innsbruck, Austria
- Denmark (2):
  - Danish Epilepsy Center, Dianalund
  - The Epilepsy Clinic, Glostrup Municipality
- France (11):
  - Centre Hospitalier d'Annecy, Annecy
  - CH Germon et Gauthier, Béthune
  - Hopital Pellegrin Tripode, Bordeaux
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital General, Dijon
  - Hopital Victor Jousselin, Dreux
  - Cabinet de neurologie, Gap
  - Hopital de la Timone Adultes, Marseille
  - Groupe hospitalier Pitie Salpetriere, Paris
  - Hopital de Font Pre, Toulon
  - CHU Bretonneau, Tours
- Germany (6):
  - Universitatsklinikum Campus Virchow-Klinikum Wedding, Berlin
  - Epilepsieklinik Tabor, Bernau B. Berlin
  - Universitat Freiburg, Freiburg im Breisgau
  - Epilepsiezentrum Kork, Kehl-Kork
  - Arzneimittelforschung Leipzig GmbH, Leipzig
  - Klinik die Weissenau, Revensburg
- Italy (8):
  - Ospedale Riuniti di Bergamo, Bergamo
  - Azienda Ospedaliero- Universitaria Policlinico di Catania, Catania
  - Istituto Nazionale Neurologico Carlo Besta di Milano, Milan
  - Azienda Ospedaliera San Paolo, Milan
  - Universita di Parma, Parma
  - Azienda Ospedaliera Bianchi-Melancrino-Morelli, Reggio Calabria
  - Universita degli studi La Sapienza, Roma
  - Universita degli Studi La Sapienza, Roma
- Norway (3):
  - Nevrologisk avdelning, 10 etasje, Lillehammer
  - Sandvika Neurologpraksis, Sandvika
  - Avd. for nevrologi og klinisk nevrofysiologi, Trondheim
- United Kingdom (2):
  - University Hospital of Wales, Cardiff
  - University Hospital of North Staffordshire Royal Infirmary, Stoke-on-Trent